CLINICAL TRIAL: NCT03589755
Title: The Impact of Mindfulness Meditation in Veterans With Epilepsy: Can Seizures and Psychiatric Comorbidities Improve
Brief Title: The Impact of Mindfulness Meditation in Veterans With Epilepsy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit enough candidates
Sponsor: Miami VA Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Maria Raquel Lopez, Primary Investigator, Miami VA Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1158499-1
Record Dates: First submitted 2018-05-14; First posted 2018-07-18 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Epilepsy
Keywords: mindfulness; meditation; anxiety; depression
MeSH Terms: conditions — Epilepsy; Anxiety Disorders; Depression | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Clinical providers in the epilepsy clinic are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mindful meditation (Active Comparator): Behavioral intervention, providing meditation
  Interventions: Behavioral: Mindfulness meditation
- Waiting list (No Intervention): Patient on a waiting list

INTERVENTIONS:
Behavioral: Mindfulness meditation — The intervention consist of a weekly session of mindfulness meditation provided by a clinical psychologist trained in this area. She will provide weekly session to a group of 10 patients at a time for a total of 8 weeks. Upon completing the course, the other 10 people will start
  Arms: mindful meditation

SUMMARY:
Epilepsy is one of the fourth most common neurological disorder and affects people of all ages and about 25 % of those patients have medically intractable epilepsy. Since the traditional pharmaceutical and surgical approach is not always effective, this study intends to investigate a novel approach using mindfulness as adjunctive tool of treatment for veterans with epilepsy.

This study proposes a randomized, single-blinded pilot investigative trial to assess the effectiveness of mindfulness meditation. The measures outcomes include seizure frequency, number of ER visits, quality of life, depression, anxiety, post traumatic stress disorder (PTSD), sleep quality and alcohol use in patients with Epilepsy. The cohort group will be randomized in two groups, one is the group of patients getting mindful meditation weekly during 8 weeks compared to patients in the waiting list who have the desire to participate.

DETAILED DESCRIPTION:
This is a randomized control trial of the impact of mindfulness meditation in patients with known diagnosis of epilepsy over the course of 2 years.

Participating physicians will recruit patients meeting the inclusion and exclusion criteria who have been diagnosed and treated in the epilepsy clinic at the Miami Veteran hospital. Upon completion of screening and enrolment procedures study participants will be randomly assigned to one of the two groups using a randomized call-in system: Treatment with weekly sessions of mindfulness meditation for 8 weeks or placement in the waiting list.

Demographics will be obtained for both groups during the initial clinic visit. The epilepsy variable questionnaire will also be completed during the initial appointment in the epilepsy clinic (this will assess seizure frequency, number of ER visits 3 months prior, adherence to antiepileptic medications reviewing the electronic pharmacy log with dates of medication being dispensed at the Veteran Medical Center.

All patients will be scheduled to have an initial appointment with the clinical psychologist to fill out the complete a battery of questionnaires including: Quality of life inventory in epilepsy (QOLIE-31), alcohol use disorder identification test (AUDIT), Beck depression inventory (BDI-II), Beck anxiety inventory (BAI), drug abuse screening test (dast-10), Epworth Sleepiness Scale, Insomnia severity, patient health questionnaires (PHQ), Post traumatic

The patients who do not initially receive mindfulness meditation will continue to receive standard of care and will be placed in a second phase of randomization where they will have a chance to once again be randomized to one of the groups.

This process will continue until a total of at least 40 patients has been recruited. After the recruitment has been completed, the remainder of the patients will be given the opportunity to participate in mindfulness medication if they so desire.

The hypothesis is that mindfulness meditation group will have more favorable outcomes than patients in the waitlist group in terms of the primary outcome of reduction in seizure frequency and secondary outcomes including number of ER visits, improvement in quality of life, decreasing symptoms of depression, anxiety, and/or PTSD, improvement in sleep quality, and decreased alcohol use.

Physicians will be blinded to which group patients are assigned during data collection. All of the participants will have a weekly clinic note titled Psychology Note in the clinic MIA MH PSYCHOL MINDFUL GRP. The notes will document the session if patient is in the mindfulness meditation group or will document that the patient remains on the waiting list. The physicians will not access these notes and will remain blinded to the patient assignment and upon completion of the study the data will be de-identified and analyzed by the statistician.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of epilepsy, according to the using the 2014 International League Against Epilepsy criteria
2. Adults over the age of 18
3. Willingness to participate in mindfulness meditation sessions weekly for 8 weeks
4. Being able to read at a 6th grade level.
5. Being able to understand the study, consent form, and guided instructions during mindfulness meditation.

Exclusion Criteria:

1. Having an isolated diagnosis of psychogenic non-epileptic seizures.
2. Having a diagnosis of major neurocognitive disorder previously known as dementia which would make the patient unable to follow guided instructions during mindfulness meditation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Change in number of seizures over time | Number of seizures in 4 weeks (baseline) prior to beginning the mindfulness study and then week 4, 8 and 12 from the begining of the study.
  Total number of seizures per 4 week periods will be compared over time.

SECONDARY OUTCOMES:
Change in number of Emergency room (ER) visits | At the beginning of study ( will iclude number of ER visit 3 month prior to enrollment in study. Then at week 12 and 3 months after completing the study.
  Number of ER visits during 3 months (baseline) prior to meditation study compared with number of ER visits during three months after the completion of meditation.
Change in quality of life in epilepsy questionnaire (QOLIE-31) scores over time | At the beginning of mindfulness study (baseline) and then at the end of weeks 4 and 8 during mindfulness study and one month after completion of meditation sessions (post study)
  Score of QOLIE - 31 at the baseline, then at week 4 and week 8 during meditation study and 4 weeks after the completion of study. The QoLIE-31 score range is from 0 to 100 with a higher score indicating a better outcome for quality of life.

OTHER OUTCOMES:
Change in beck depression inventory I and II (BDI-II) scores over time | baseline scores at the beginning of study, at the end of week 4 and week 8 during mindfulness study and a month after completing the study (at the end of week 12)
  We will compare the scores of BDI-II at the baseline, and after week 4 and week 8 during meditation study and 4 weeks after the completion of study. The BDI-II score range is from 0 to 63 with a higher score indicating a worsening of depression.
Change in the Beck anxiety inventory (BAI) scores over time | At the beginning of mindfulness study (baseline) and then at the end of weeks 4 and 8 during mindfulness study and one month after completion of meditation sessions (post study)
  We will compare the scores of the DAI at the baseline, then at the end of week 4 and week 8 during meditation study and 4 weeks after the completion of study. The BAI score range is from 0 to 63 with a higher score indicating a worsening anxiety.
Change in the drug abuse screening test (dast-10) scores over time | At the beginning of mindfulness study (baseline) and then at the end of weeks 4 and 8 during mindfulness study and one month after completion of meditation sessions (post study)
  We will compare the scores of the dast-10 at the baseline, then at the end of week 4 and week 8 during the meditation study and a month after the completion of the study. The dast 10 score range from 0 to 10 with a higher number indicating a worse drug addiction.
Change in the Epworth Sleepiness Scale (ESS) | At the beginning of mindfulness study (baseline) and then at the end of weeks 4 and 8 during mindfulness study and one month after completion of meditation sessions (post study)
  We will compare the score of the ESS at the baseline, then 4, 8 and 12 week after the baseline testing. The ESS score range is from 0 to 24 with a higher score indicating higher chance of dozing
Change in the Alcohol use disorder identification test (AUDIT) | At the beginning of mindfulness study (baseline) and then at the end of weeks 4 and 8 during mindfulness study and one month after completion of meditation sessions (post study)
  Score of AUDIT at the baseline, then at week 4 and week 8 during meditation study and 4 weeks after the completion of study. The AUDIT score range from 0 to more than 20 with a higher score indicating a higher use of alcohol
Change of the insomnia severity index score (ISIS) | At the beginning of mindfulness study (baseline) and then at the end of weeks 4 and 8 during mindfulness study and one month after completion of meditation sessions (post study)
  We will compare the score of ISIS at baseline, then at week 4 and week 8 during meditation study and 4 weeks after the completion of the study. The ISIS score range is from 0 to 28 with a higher score indicating higher severity of insomnia
Change of the patients health questionnaire (PHQ-9) score | At the beginning of mindfulness study (baseline) and then at the end of weeks 4 and 8 during mindfulness study and one month after completion of meditation sessions (post study)
  Score of PHQ questionnaire at the baseline, then at week 4 and week 8 during meditation study and 4 weeks after the completion of study. The PHQ-9 score range is from 0 to 27 with a higher score indicating a more severe depression.
Change of the PCL-5 scores | At the beginning of mindfulness study (baseline) and then at the end of weeks 4 and 8 during mindfulness study and one month after completion of meditation sessions (post study)
  The PCL- 5 is a 20-item self report measure that assesses the 20 DSM-5 symptoms of the PTSD .We will compare the scores of the PCL-5 at the baseline, then at the end of week 4 and week 8 during the meditation study and 4 weeks after the completion of the study. PCL for DSM-IV suggests that a 5-10 point change represents reliable change (i.e., change not due to chance) and a 10-20 point change represents clinically significant change.

CONTACTS AND LOCATIONS:
Overall Officials: Maria R Lopez, M.D, Principal Investigator — Miami Veteran Affairs hospital
Locations (1):
- miami VAMC, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access request will be reviewed by an external independent reviewer panel. Requests will be required to sign a data access agreement
URL: http://IRBNET.org

REFERENCES:
- [Result] Hauser WA, Annegers JF, Rocca WA. Descriptive epidemiology of epilepsy: contributions of population-based studies from Rochester, Minnesota. Mayo Clin Proc. 1996 Jun;71(6):576-86. doi: 10.4065/71.6.576. PMID 8642887
- [Result] Arias AJ, Steinberg K, Banga A, Trestman RL. Systematic review of the efficacy of meditation techniques as treatments for medical illness. J Altern Complement Med. 2006 Oct;12(8):817-32. doi: 10.1089/acm.2006.12.817. PMID 17034289
- [Result] Vezzani A, Lang B, Aronica E. Immunity and Inflammation in Epilepsy. Cold Spring Harb Perspect Med. 2015 Dec 18;6(2):a022699. doi: 10.1101/cshperspect.a022699. PMID 26684336
- [Result] Pascoe MC, Thompson DR, Jenkins ZM, Ski CF. Mindfulness mediates the physiological markers of stress: Systematic review and meta-analysis. J Psychiatr Res. 2017 Dec;95:156-178. doi: 10.1016/j.jpsychires.2017.08.004. Epub 2017 Aug 23. PMID 28863392
- [Result] Walker ER, Obolensky N, Dini S, Thompson NJ. Formative and process evaluations of a cognitive-behavioral therapy and mindfulness intervention for people with epilepsy and depression. Epilepsy Behav. 2010 Nov;19(3):239-46. doi: 10.1016/j.yebeh.2010.07.032. Epub 2010 Sep 15. PMID 20833592
- [Result] Acevedo BP, Pospos S, Lavretsky H. The Neural Mechanisms of Meditative Practices: Novel Approaches for Healthy Aging. Curr Behav Neurosci Rep. 2016;3(4):328-339. doi: 10.1007/s40473-016-0098-x. Epub 2016 Oct 18. PMID 27909646
- [Result] Moyer CA, Donnelly MP, Anderson JC, Valek KC, Huckaby SJ, Wiederholt DA, Doty RL, Rehlinger AS, Rice BL. Frontal electroencephalographic asymmetry associated with positive emotion is produced by very brief meditation training. Psychol Sci. 2011 Oct;22(10):1277-9. doi: 10.1177/0956797611418985. Epub 2011 Sep 15. No abstract available. PMID 21921291
- [Result] Tang YY, Lu Q, Feng H, Tang R, Posner MI. Short-term meditation increases blood flow in anterior cingulate cortex and insula. Front Psychol. 2015 Feb 26;6:212. doi: 10.3389/fpsyg.2015.00212. eCollection 2015. PMID 25767459
- [Result] Guidelines for epidemiologic studies on epilepsy. Commission on Epidemiology and Prognosis, International League Against Epilepsy. Epilepsia. 1993 Jul-Aug;34(4):592-6. doi: 10.1111/j.1528-1157.1993.tb00433.x. No abstract available. PMID 8330566